CLINICAL TRIAL: NCT04766437
Title: Optical Coherence Tomography-Guided PCI With Single-Antiplatelet Therapy
Acronym: OPTICA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPTICA
Record Dates: First submitted 2021-02-18; First posted 2021-02-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Non ST Segment Elevation Acute Coronary Syndrome
Keywords: Non ST Segment Elevation Acute Coronary Syndrome; Percutaneous coronary intervention; Prasugrel monotherapy; Ticagrelor monotherapy; P2Y12-inhibitor monotherapy
MeSH Terms: interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Intervention Model Description: Single arm pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prasugrel or ticagrelor monotherapy (Experimental): Once daily 10 mg prasugrel or twice daily 90 mg ticagrelor for 12 months preceded by a loading dose of 60 mg prasugrel or 180 mg ticagrelor at least 2 hours prior to percutaneous coronary intervention without concurrent aspirin therapy.
  Interventions: Drug: Prasugrel 10mg; Drug: Ticagrelor 90mg

INTERVENTIONS:
Drug: Prasugrel 10mg — Once daily 10 mg prasugrel for 12 months preceded by a loading dose of 60 mg prasugrel at least 2 hours prior to percutaneous coronary intervention without concurrent aspirin therapy.
Drug: Ticagrelor 90mg — Twice daily 90 mg ticagrelor for 12 months preceded by a loading dose of 180 mg ticagrelor at least 2 hours prior to percutaneous coronary intervention without concurrent aspirin therapy.

SUMMARY:
Rationale: Dual antiplatelet therapy, consisting of aspirin and a P2Y12-inhibitor, reduces the risk of stent thrombosis, myocardial infarction and stroke after coronary stent implantation. Inevitably, it is also associated with a higher risk of (major) bleeding. Given the advances in stent properties, stenting implantation technique and pharmacology, it may be possible to treat patients with a single antiplatelet strategy using a potent P2Y12-inhibitor such as prasugrel or ticagrelor.

Objective: This study will serve as a pilot to investigate the feasibility and safety of a single antiplatelet strategy with prasugrel or ticagrelor prior to, during and after stent implantation in 75 patients with non-ST segment elevation acute coronary syndrome.

Study design: Single-center, single arm pilot study with a stopping rule based on the occurrence of definite stent thrombosis.

Study population: Patients presenting with non-ST segment elevation acute coronary syndrome and (a) 'de novo' lesion(s) treated with new generation drug-eluting stent(s) with adequate reduction of platelet reactivity according to platelet function testing with VerifyNow and optimal stenting result adjudicated by optical coherence tomography or coronary angiography.

Intervention: Once daily 10 mg prasugrel or twice daily 90 mg ticagrelor for 12 months preceded by a loading dose of 60 mg prasugrel or 180 mg ticagrelor at least 2 hours prior to percutaneous coronary intervention without concurrent aspirin therapy.

Main study endpoint: The primary ischemic endpoints is the composite of all-cause mortality, myocardial infarction, Academic Research Consortium defined stent thrombosis and ischemic stroke at 6 months after percutaneous coronary intervention. The primary bleeding outcome is major or minor bleeding defined as Bleeding Academic Research Consortium type 2, 3 or 5 bleeding at 6 months after percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* NSTE-ACS diagnosis
* 'De novo' coronary lesion(s) eligible for PCI
* Written informed consent

Exclusion Criteria:

* Known allergy or contraindication for prasugrel and ticagrelor use.
* Concurrent use of oral anticoagulants
* Overwriting indication for DAPT
* Planned surgical intervention within 12 months of planned revascularization
* PCI of left main disease, chronic total occlusion, bifurcation lesion requiring two-stent treatment, saphenous or arterial graft lesion, severely calcified lesions
* Recent or ongoing strong CYP3A4 inhibitor or inducer therapy
* Recent or ongoing therapy with CYP4A4-substrates with a narrow therapeutic index
* Pregnant or breastfeeding women at time of enrolment
* Participation in another trial with an investigational drug or device (i.e. stent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2022-09-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Primary ischemic endpoint | 6 months
  Number of participants with primary ischemic endpoint defined as composite of all-cause mortality, myocardial infarction, Academic Research Consortium defined stent thrombosis and ischemic stroke
Primary bleeding endpoint | 6 months
  Number of participants with primary bleeding endpoint defined as Bleeding Academic Research Consortium type 2, 3 or 5 bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided